CLINICAL TRIAL: NCT01153984
Title: Biomarkers Impact on the Response to Treatment With Erlotinib in First Line Non-small Cell Lung Cancer With EGFR Activating Mutations - BIOTEC
Brief Title: A Study to Assess Biomarkers Impact on Participants Response to Erlotinib Treatment for First-line Non-Small Cell Lung Cancer With Endothelial Growth Factor Receptor (EGFR) Activating Mutations
Acronym: BIOTEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22606; 2009-017063-42
Record Dates: First submitted 2010-06-16; First posted 2010-06-30 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma，Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib (Experimental): Participants will receive 150 milligrams (mg) erlotinib orally daily until disease progression, unacceptable toxicity, withdrawal due to any reason or death.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150 mg oral doses will be administered daily.
  Other Names: Tarceva

SUMMARY:
This open-label, single-arm, multi-center study will evaluate the progression-free survival in participants with histologically documented, advanced and/or metastatic chemotherapy naive, non-small cell lung cancer (NSCLC) with Epidermal Growth Factor Receptor (EGFR) positive mutations and receiving erlotinib treatment. The anticipated time on study treatment is until disease progression, unacceptable toxicity, withdrawal due to any reason or death.

ELIGIBILITY:
Inclusion Criteria:

* Histological documented adenocarcinoma, locally advanced - Stage IIIB, metastatic - Stage IV or recurrent non-squamous NSCLC
* Activated EGFR mutation positive status (Exons 19 and 21) for treatment phase
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy greater than or equal to (≥) 12 weeks
* Evidence of disease with at least one measurable disease evaluation on Response Evaluation Criteria in Solid Tumors (RECIST)
* Adequate hematological , liver and renal function

Exclusion Criteria:

* Known hypersensitivity to erlotinib or any of its excipients
* Squamous non-small cell or small cell tumors or absence of histological report
* Neoadjuvant/adjuvant chemotherapy within 6 months prior to enrollment
* Prior exposure to inhibitors of EGFR
* Prior chemotherapy or treatment with another systemic anti-cancer agent for the treatment of the participant's current stage of disease
* Any significant ophthalmologic abnormality, especially severe dry eye syndrome, keratoconjunctivitis sicca, Sjögren syndrome, severe exposure keratitis or any other disorder likely to increase the risk of corneal epithelial lesions
* Radical radiotherapy with curative intent within 28 days prior to enrollment
* Any active non-controlled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Romania (9):
  - County Hospital Alba; Oncology, Alba Iulia
  - Institut of Oncology Al. Trestioreanu Bucharest; Oncology, Bucharest
  - Institute Of Oncology Bucharest; Medical Oncology, Bucharest
  - Spitalul de Boli Cronice Sf. Luca, Bucharest
  - Emergency University Bucharest Hospital; Oncology Department, Bucharest
  - Oncology Inst. Cluj-Napoca; Cancer Dept, Cluj-Napoca
  - Uni Hospital St. Spiridon; Clinica Oncologie-Radiotherapie, Iași
  - S.C. Life Search S.R.L; Medical Oncology Clinic, Timișoara
  - ONCOMED - Medical Centre, Timișoara

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ninety participants were screened and 23 participants were enrolled.
Groups:
- Erlotinib: Participants received 150 milligrams (mg) erlotinib orally daily until disease progression, unacceptable toxicity, withdrawal due to any reason or death.
Period: Overall Study
Arm/Group | Erlotinib
Started | 23
Completed | 21
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants.
Groups:
- Erlotinib: Participants received 150 mg erlotinib orally daily until disease progression, unacceptable toxicity, withdrawal due to any reason or death.
Arm/Group | Erlotinib
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.52 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS), as Assessed by Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: PFS was the time from inclusion in the study to the date of first documented PD or death from any cause, whichever occurred first. Participants without event were censored at the date of the last tumor assessment where non-progression was documented. If a participant received a second anti-cancer therapy without prior documentation of disease progression, the participant was censored at the date of last tumor assessment before starting new chemotherapy. Analysis was performed using Kaplan-Meier method. PD was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: Baseline up to approximately 4 years
Population: All enrolled participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib
Number analyzed (Participants) | 23
days | 387.000 (85.32) [103.592 to 670.408]

2. Secondary Outcome: Time to Disease Progression, as Assessed by Investigator Using RECIST v1.1
Description: Time to disease progression was defined as the time from baseline evaluation to the first date PD was recorded. Participants without progression were censored at the date of last tumor assessment where non-progression was documented. PD was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: Baseline up to approximately 4 years
Population: All enrolled participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib
Number analyzed (Participants) | 23
days | 193.00 (70.323) [57.137 to 328.863]

3. Secondary Outcome: Percentage of Participants With Complete Response (CR) And Partial Response (PR) as Assessed by the Investigator Using RECIST v1.1
Description: CR was defined as the disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of the longest diameter compared to baseline.
Time Frame: Baseline up to approximately 4 years
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 23
percentage of participants
  CR | 0
  PR | 8.7

4. Secondary Outcome: Percentage of Participants Who Were Alive One Year After Study Treatment Initiation
Time Frame: Year 1
Population: All enrolled participants with available data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 21
percentage of participants | 85.7

5. Secondary Outcome: Percentage of Participants by Localization of PD, as Assessed by Investigator Using RECIST v1.1
Description: PD was assessed using RECIST v1.1. PD was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. Percentage of participants by localization of PD were reported. Localization included: Left lung inferior lobe; Para-aortic; Left lung upper lobe; Right lung inferior lobe; and Infracranial.
Time Frame: Baseline up to approximately 4 years
Population: All enrolled participants with available data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 21
percentage of participants
  Left lung inferior lobe | 24
  Para-aortic | 14
  Left lung upper lobe | 10
  Right lung inferior lobe | 14
  Infracranial | 38

6. Secondary Outcome: Number of EGFR Positive Participants Classified Based on Smoking Status
Description: Participants were asked: "Have you smoked at least 100 cigarettes in your entire life?" and "Do you now smoke cigarettes every day, some days, or not at all?" Responses were grouped into three categories: Current Smoker, Former Smoker, and Non-Smoker. Participants who reported smoking at least 100 cigarettes in their lifetime and who, at the time of survey, smoked either every day or some days were defined as 'Current smoker'. Participants who reported smoking at least 100 cigarettes in their lifetime and who, at the time of the survey, did not smoke at all were defined as 'Former smoker'. Participants who reported never having smoked 100 cigarettes were defined as 'Non-smoker'.
Time Frame: Day 1
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 23
participants
  Non-smoker | 17
  Former smoker | 3
  Current smoker | 3

7. Secondary Outcome: Number of EGFR Positive Participants Classified Based on Type of EGFR Mutations
Description: Participants with NSCLC have tumor associated with EGFR mutations. These mutations occur within EGFR Exons 18-21, which encodes a portion of the EGFR kinase domain.
Time Frame: Day 1
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 23
participants
  Exon 19 deletions | 20
  Exon 21 L858R mutations | 3

8. Secondary Outcome: Percentage of Similar EGFR Mutations Between Matched Plasma and Tumor Tissue Samples
Time Frame: Baseline up to approximately 4 years
Population: No participants were analyzed for this outcome as no plasma samples were collected during the study.
Arm/Group | Erlotinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 4 years
Description: Safety analysis population included all participants who receive at least one dose of treatment and had at least one monthly assessment.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 5/23
Other Adverse Events (participants affected / at risk) | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=23)
Hemiparesis (Nervous system disorders) | 1
Brain neoplasm malignant (Nervous system disorders) | 1
Respiratory tract infection (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Ischemic stroke (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=23)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vomiting (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Vaginal hemorrhages (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 8
Chest pain (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Transaminases increased (Investigations) | 1
Rash (Skin and subcutaneous tissue disorders) | 7
Conjunctivitis (Eye disorders) | 1
Syncope (Cardiac disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Menorrhagia (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.